CLINICAL TRIAL: NCT04812613
Title: Tobacco Concurrent Addictions in At-Risk Youth in Ottawa: A Mixed Methods Community-Based Participatory Action Research Project (TCAY- Ottawa)
Brief Title: Tobacco-Concurrent Addictions in At-Risk Youth in Ottawa
Acronym: TCAY-Ottawa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Operation Come Home (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20180595-01H
Record Dates: First submitted 2019-12-11; First posted 2021-03-23 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Tobacco Use; Substance Use
MeSH Terms: conditions — Tobacco Use; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Photovoice: Three youth community peer researchers from marginalized communities will be recruited and involved in every aspect of the project.
  We will recruit 20 participants from marginalized communities with a current or past history of cannabis use, who can speak English, and who are between 16 and 26 years old.
  Participants will receive training on study procedures, basics of photography and disposable camera to document their experiences with mental health and substance use over the span of two weeks. Community peer researchers and research team will conduct photoanalysis and creation of the description of the five photos chosen by each participant.
  Duoethnographic dialogue: 10 youth participants will be paired with an older participant of TCAY study to have an open discussion to explore their experiences with cannabis and mental health. This conversation will be facilitated by community peer researcher, recorded and transcribed verbatim.
- Mix-method community based participatory action research: Phase 1 study: we will conduct 50 semi-structured questionnaires. Data from the participants and literature will then be triangulated, coded, and analyzed using NVivo software. Researchers will transcribe interviews, create a code guide, code, analyze and report the data to appropriately inform the intervention (Phase 2).
  Phase 2: 6 month follow-up with a questionnaire focused on socio-demographic data, questions on participants' smoking and other substance use habits, mental health, as well as questions on participants' social networks.. Participants will be informed that they can skip any of the questions if they are uncomfortable answering them. Qualitative data will be analyzed using NVivo, and quantitative data will be analyzed using SAS or R software. Phase 2 findings will be reported and submitted to an appropriate peer-review journal.

SUMMARY:
According to the 2015 Ontario Student Drug Use and Health Survey (OSDUHS), there has been a significant increase in the number of secondary school youth who use poly-substances. Not all youth have the same risk for problematic substance use. Health literature documents a high level of comorbidity between mental health and substance use, which is exacerbated in homeless youth populations. Therefore, the proposed study will focus on understanding poly-substance use among at-risk homeless school youth. As seen in substance use research and the PROMPT (2016) study (Participatory Research in Ottawa: Management and Point-of-Care for Tobacco Dependence, PI: Dr. Smita Pakhale), reduction and quitting of one substance (tobacco smoking) can lead to the reduction and quitting of other poly-substance use. A Community-Based Participatory Action Research (CBPAR) approach can help at-risk youth feel safe and comfortable enough to provide personal information about their poly-substance use and engagement with treatment or harm reduction programs. This project will be a first step in increasing health equity among at-risk homeless youth in Downtown Ottawa. The investigators aim to follow a group of at-risk youth to while providing an appropriately modified PROMPT intervention, including peers support and a licensed mental health and substance use nurse.

DETAILED DESCRIPTION:
Research Objectives:

Understand the real reasons that impact cannabis use, positive and negative experiences for that, how much cannabis use effect on mental health, recognize the patterns of cannabis use between deferent generation among marginalized populations with a disproportionate burden of mental illness. Also, use meaningful qualitative method to encourage storytelling and authentic sharing of individual experiences of mental health and cannabis use.

Primary Patient-Oriented Outcome: Improved engagement and quality of life in participants. As well, reduced self-reported poly-substance use.

Study Design: Phase 1: will involve gathering information on the root causes or facilitators of poly-substance use among at-risk youth, the types of drug use that is most prevalent among at-risk youth, and the early and ongoing points of access to licit and illicit substances. Phase II: will involve a single arm prospective cohort study looking to tackle poly-substance use in marginalized youth by providing an individualized, youth-tailored (i.e. based on qualitative results obtained in phase I), social-based intervention with optional access to an licensed mental health and substance use nurse counselling. Photovoice: The 20 recruited participants will be trained on how to use Photovoice. Dialogue: Ten interested Photovoice participants will be invited to be paired one-on-one with an adult-aged (aged 27+) participant of the MHCC OCM project.

Setting: 1) The Bridge Engagement Centre, Ottawa and 2) Operation Come Home, Ottawa

Expertise: The PI is well versed in community-based research. Dr. Pakhale led the PROMPT project, a community-based smoking cessation project engaging a similar target population. Partnering with Operation Come Home and Ms. Elspeth McKay, the executive director of Operation Come Home, provides the PI with expert experience in engaging this marginalized youth population. Together the team is very experienced in substance dependence and the target population. The investigators collective expertise with links to the target community will support the implementation of the trial.

Outcomes: Community-based participatory and peer-led research holds a tremendous potential in investigating solutions 'for the people, by and with the people'. Outcomes of this trial will aid policy makers in designing and implementing effective programs to treat substance dependence in marginalized youth populations.

Timeline: Participants will be invited to complete the study-specific survey monthly, for 6-months.

ELIGIBILITY:
Inclusion criteria:

* Are currently living in Ottawa for at least 3 months prior to enrolment.
* Are homeless or insecurely housed (from OCH and the Bridge).
* 16 years or older.
* currently use or have a past history of cannabis use
* Self-report a mental illness.

Exclusion criteria:

• Not meeting inclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 20 youth and 200 adult participants
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Explore the frequency of tobacco and other drug use | 6 Months
  Understand the problem of substance use and addiction among youth between the ages of 16 years or older who are homeless or insecurely housed (as defined-by project step) in Downtown Ottawa, and who attend programs at project step partner, OCH
Tobacco and other drug use reduction | 6 Months
  Design and deliver an individualized intervention (6 months) to help at-risk youth decrease concurrent poly-substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Pakhale, M.D., Principal Investigator — Ottawa Hospital
Locations (1):
- The Bridge Engagement Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes